CLINICAL TRIAL: NCT00436462
Title: Expression of Steroid Receptors in Endometrium During the Early Follicular Phase in Stimulated Cycles
Brief Title: Expression of Steroid Receptors in Endometrium
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Unit for Human Reproduction, Aristotle University of Thessaloniki
Other Study IDs: UHR-4
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Endometrium
Keywords: Steroid receptors; Endometrium; IVF; Follicular phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — endometrial tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Expression of steroid receptors in endometrium during ovarian stimulation.

DETAILED DESCRIPTION:
The purpose of this study is to examine in stimulated cycles a) whether there is a difference in expression of steroid receptors in stroma and glands of endometrium between different days during the follicular phase b)whether there are secretory changes detected by endometrium histology before ovulation c)whether there is an association between expression of steroid receptors in endometrium and exposure to oestradiol and progesterone during the follicular phase.

ELIGIBILITY:
Inclusion Criteria:

* Treatment by IUI,
* BMI:18-29KGR/M2,
* No previous ovarian surgery,
* Normal hysterosalpingography,
* Estradiol < 80pg/ml and progesterone < 1.6ng/ml on day 2 of the cycle

Exclusion Criteria:

* Endometriosis,
* Severe male factor

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: infertile women
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Steroid receptors expression in endometrium during early follicular phase | 3 months

SECONDARY OUTCOMES:
In which day:day o+2, day 0+4 or day HCG | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Basil C Tarlatzis, MD,PhD, Study Director — Unit of Human Reproduction, 1st Department of Obst & Gyn, Aristotle University of Thessaloniki, Papageorgiou Hospital, Greece
Locations (1):
- Unit of Human Reproduction, 1st Department of Obstetrics & Gynecology, AUTH, Papageorgiou Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Kolibianakis E, Bourgain C, Albano C, Osmanagaoglu K, Smitz J, Van Steirteghem A, Devroey P. Effect of ovarian stimulation with recombinant follicle-stimulating hormone, gonadotropin releasing hormone antagonists, and human chorionic gonadotropin on endometrial maturation on the day of oocyte pick-up. Fertil Steril. 2002 Nov;78(5):1025-9. doi: 10.1016/s0015-0282(02)03323-x. PMID 12413988
- [Background] Papanikolaou EG, Bourgain C, Kolibianakis E, Tournaye H, Devroey P. Steroid receptor expression in late follicular phase endometrium in GnRH antagonist IVF cycles is already altered, indicating initiation of early luteal phase transformation in the absence of secretory changes. Hum Reprod. 2005 Jun;20(6):1541-7. doi: 10.1093/humrep/deh793. Epub 2005 Feb 10. PMID 15705618